CLINICAL TRIAL: NCT00779909
Title: Dose-dependent Anti-inflammatory Effects of Vitamin D in a Human Gingivitis Model
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-26461; R21AT003714-01 (NIH)
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-08

CONDITIONS: Gingivitis
Keywords: vitamin D; gingivitis; periodontal disease; inflammation
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Inflammation | interventions — Cholecalciferol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1- Placebo (Placebo Comparator): placebo capsule once per day
  Interventions: Other: Placebo
- 2- Vitamin D3, 500 IU (Experimental): vitamin D3, 500 IU capsule once per day
  Interventions: Drug: vitamin D3
- 3- Vitamin D3, 2500 IU (Experimental): vitamin D3, 2500 IU capsule once per day
  Interventions: Drug: vitamin D3
- 4- Vitamin D3, 5000 IU (Experimental): vitamin D3, 5000 IU capsule once per day
  Interventions: Drug: vitamin D3

INTERVENTIONS:
Drug: vitamin D3 — oral supplementation once per day for 12 weeks of different daily doses: 500 IU, 2500 IU, or 5000 IU after abstaining from oral hygiene measures (brushing, flossing or antiseptic mouth rinses) for a period of 4 weeks to allow accumulation of plaque and development of experimental gingivitis.
  Other Names: cholecalciferol
  Arms: 2- Vitamin D3, 500 IU; 3- Vitamin D3, 2500 IU; 4- Vitamin D3, 5000 IU
Other: Placebo — oral supplementation once per day for 12 weeks of a sugar pill after abstaining from oral hygiene measures (brushing, flossing or antiseptic mouth rinses) for a period of 4 weeks to allow accumulation of plaque and development of experimental gingivitis.
  Other Names: sugar pill
  Arms: 1- Placebo

SUMMARY:
The burden of chronic gingivitis and periodontitis in the US is disproportionately high among Non-Hispanic Blacks compared to Non-Hispanic Whites. Chronic gingivitis is a highly prevalent chronic inflammatory disease that may progress into periodontitis, a major cause of tooth loss, Data from in-vitro and animal studies suggest anti-inflammatory effects of vitamin D; however, if and over what dose-range vitamin D may have anti-inflammatory effects in humans is uncertain. Recent clinical studies indicate that beneficial effects of vitamin D for several important outcomes may occur over a wide range of serum 25-hydroxyvitamin D (25-OHD) concentrations, possibly up to concentrations that would require vitamin D intakes ranging from 2 to more than 10 ten times higher than the current RDA for vitamin D. Because dark skin pigmentation is a potent inhibitor of vitamin D photosynthesis, Non-Hispanic Blacks have much lower 25-OHD serum levels than Non-Hispanic Whites. These differences in vitamin D status may partially explain the racial disparities in prevalence of chronic gingivitis and periodontitis observed in the US.

We hypothesize that oral cholecalciferol supplementation can reduce susceptibility to gingivitis over a wide range of serum 25-OHD concentrations in Non-Hispanic Whites and Non-Hispanic Blacks. We propose to conduct a simple, single-center, randomized, double-blind, placebo-controlled parallel-group dose-ranging study. We will compare placebo to doses of 500 IU, 2,500 IU and 5,000 IU vitamin D3 per day. We will compare the severity of gingival inflammation that develops in response to a 28-day period of unlimited plaque growth (experimental gingivitis) between dosage groups. Furthermore, we will evaluate the association between achieved 25-OHD levels and gingival inflammation.

The results of this study will have several important implications, as dietary vitamin D supplementation may be a simple, safe and inexpensive means by which to reduce racial/ethnic disparities in gingivitis, as well as to reduce the overall burden of oral disease in the population as a whole. The study will elucidate the dose-response relationship of the anti-inflammatory effects of vitamin D, which in turn may lead to a revision of the current recommendations regarding nutritional supplementation of vitamin D in order to optimize the prevention of important medical conditions and diseases and reduce racial health disparities.

DETAILED DESCRIPTION:
Vitamin D is important for healthy bones. More recently, anti-inflammatory effects of vitamin D have been found in laboratory and animal studies and vitamin D may be beneficial for inflammatory diseases. Gingivitis is a common inflammatory disease of the gums that develops in response to bacterial components in dental plaque. The degree to which gingivitis develops in response to a given amount of plaque may vary between different individuals. With this study, we want to investigate whether oral supplementation with vitamin D can reduce the susceptibility to gingivitis in non-Hispanic Whites and African Americans.

We plan to randomize 120 healthy volunteers (60 Non-Hispanic Whites, 60 Non-Hispanic Blacks) during the wintertime who will abstain from oral hygiene measures (brushing, flossing or antiseptic mouth rinses) for a period of 4 weeks to allow accumulation of plaque and development of gingivitis. These subjects will be randomly allocated to receive either oral supplementation with placebo, 500 IU, 2500 IU or 5000 IU vitamin D3 per day starting 8 weeks prior to the experimental gingivitis period for a total of 12 weeks. The development of gingivitis will be measured using clinical indices of gingival inflammation, inflammatory biomarker in gingival crevicular fluid (GCF) and GCF volume. Before and after completion of the experimental gingivitis phase, all subjects will receive a professional cleaning of their teeth to ensure complete resolution of inflammation.Blood samples will be collected at the screening examination, baseline, week 7, and after week 12 (end of trial) to determine serum levels of 25-hydroxyvitamin D, parathyroid hormone , serum calcium and to archive serum and plasma samples. In addition urine samples will be collected at baseline and weeks 4,7 and 12 to determine calcium excretion and to archive urine samples for future analyses. Mandibular and maxillary Modified Gingival Index (MGI) Scores, Plaque Index (PI) scores, and GCF sampling to measure volume and assess for biomarkers (TNF-LPH, IL-1 beta, IL-2, IL-12) will be done at 8 and 12 weeks.

Following recruitment and consent those subjects deemed eligible for further screening will then be referred to the BUMC GCRC in order to have two components of the screening procedure performed:Electrocardiogram and a blood draw to be sent to Quest for analysis of Vit D and PTH levels.

The extent to which gingivitis develops during the 4-week period of plaque accumulation will be compared between the two experimental groups. Furthermore, we will evaluate the association between serum levels of 25-OHD and the development of gingivitis as well as serum markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* healthy subjects age 18-64 years old
* serum 25-hydroxyvitamin D concentration <62.5 nmol/L (<25 ng/mL)

Exclusion Criteria:

* increased risk for infectious endocarditis that require antibiotic prophylaxis prior to periodontal probing
* women who are postmenopausal
* pregnancy or planned pregnancy within the period of the trial
* Periodontitis (attachment loss ≥4 mm and probing depths≥5 mm on at least one interproximal site)
* Any need for immediate dental treatment (can be eligible after completion of treatment)
* history of hypercalcemia, malabsorption syndrome, abnormal sensitivity to vitamin D or hypervitaminosis D
* < 3 teeth with bleeding on probing
* < 20 teeth present or <8 interproximal spaces (i.e., papillae) in upper jaw
* mean plaque index > 3
* Current smoking or former smoking with cessation <5 years ago
* regular use of any medication for prevention or treatment of disease (including Aspirin, NSAIDs, corticosteroids, but NOT including contraceptives)
* Diabetes mellitus
* hypercalcemia (serum calcium > ULN),
* hypocalcemia (serum calcium < ULN),
* hyperparathyroidism (serum PTH concentration > ULN),
* hypoparathyroidism (serum PTH concentration < LLN)
* any cardiac rhythm abnormalities on baseline ECG
* use of tanning beds/unwillingness to abstain from use of tanning beds during study
* planned travel during study period / unwillingness to abstain from travel to the South or High Altitudes
* unwillingness to abstain from use of any supplements (including vitamin/mineral and herbal supplements) during study period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul I Garcia, DMD, Principal Investigator — Boston University School of Dental Medicine
Locations (1):
- Boston University Goldman School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 102 potential participants were screened for study eligibility, 61 met various exclusions criteria, and 41 were found to be eligible for randomization. Of the 41 eligible subjects 35 were randomized into the trial. The 6 not randomized were either lost to follow-up or they lost interest and withdrew their consent for further involvement.
Groups:
- 1- Placebo: placebo oral supplementation once per day for 12 weeks
- 2- Vitamin D3, 500 IU: vitamin D3 500 IU oral supplementation once per day for 12 weeks
- 3- Vitamin D3 2500 IU: vitamin D3 2500 IU oral supplementation once per day for 12 weeks
- 4- Vitamin D3 5000 IU: vitamin D3 5000 IU oral supplementation once per day for 12 weeks
Period: Overall Study
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
Started | 10 | 9 | 8 | 8
Completed | 9 | 8 | 8 | 7
Not Completed | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1-Placebo: placebo oral supplementation once per day for 12 weeks
- 2-Vitamin D3, 500 IU: vitamin D3 500 IU oral supplementation once per day for 12 weeks
- 3-Vitamin D3, 2500 IU: vitamin D3 2500 IU oral supplementation once per day for 12 weeks
- 4-Vitamin D3, 5000 IU: vitamin D3 5000 IU oral supplementation once per day for 12 weeks
- Total: Total of all reporting groups
Arm/Group | 1-Placebo | 2-Vitamin D3, 500 IU | 3-Vitamin D3, 2500 IU | 4-Vitamin D3, 5000 IU | Total
Number analyzed (Participants) | 10 | 9 | 8 | 8 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 8 | 8 | 35
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 7 | 5 | 23
  Male | 5 | 3 | 1 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic Black | 5 | 5 | 4 | 5 | 19
  Non-Hispanic White | 5 | 4 | 4 | 3 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 8 | 8 | 35

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Sites That Bleed on Probing
Description: Assessment of the bleeding index will be performed on oral and buccal sites. The periodontal probe will be moved gently across the marginal gingiva of all teeth of a quadrant. After 30 seconds, absence or presence of bleeding will be scored. The number of bleeding sites is used to calculate the gingival bleeding score.
Time Frame: end of 4 week experimental gingivitis phase
Population: Data for this outcome measure was not collected on any of the participants as it was overlooked and failure to collect these data did not come to the attention of the PI until after all follow-ups were completed.
Groups:
- 2- Vitamin D3, 500 IU; 3.Vitamin D3, 2500 IU; 4- Vitamin D3 5000 IU: vitamin D3: oral supplementation once per day for 12 weeks
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3.Vitamin D3, 2500 IU | 4- Vitamin D3 5000 IU
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Mandibular Modified Gingival Index (MGI) Score
Description: The Modified Gingival Index (MGI) uses non-invasive/no probing and rates mild and moderate inflammation where: 0 = absence of inflammation; 1 = mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary; 2 = mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary; 3 = moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary; 4 = severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration. The MGI can be obtained by adding the values of each tooth and dividing by the number of teeth examined. The MGI may be scored for all surfaces of all or selected teeth or for selected areas of all or selected teeth. A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation.
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
units on a scale
  8wk mandibular MGI score | 1.83 (0.27) | 1.76 (0.46) | 1.62 (0.44) | 1.67 (0.28)
  12wk mandibular MGI score | 2.12 (0.14) | 1.97 (0.24) | 2.02 (0.20) | 2.19 (0.15)

3. Primary Outcome: Maxillary Modified Gingival Index (MGI) Score
Description: as for outcome 2
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
units on a scale
  8wk maxillary MGI score | 1.78 (0.29) | 1.63 (0.40) | 1.57 (0.39) | 1.61 (0.31)
  12wk maxillary MGI score | 2.11 (0.16) | 1.87 (0.30) | 1.9 (0.30) | 2.1 (0.10)

4. Secondary Outcome: Mandibular Plaque Index (PI) Score
Description: The Turesky plaque index was used. In this index, plaque is identified using a disclosing solution and scored using a 0 to 5 scale in which a score of 0= No plaque, 1= Separate flecks of plaque, 2= continuous band of plaque less or equal 1 mm, 3= Continuous band of plaque greater than 1 mm but less than 1/3 of crown height, 4= Continuous band of plaque greater or equal 1/3 but less or equal 2/3 of crown height, and 5= Continuous band of plaque greater 2/3 of crown height. Each tooth receives 6 individual scores at: mesial, middle, and distal scores for both the facial and lingual surfaces. An individual's score is derived by adding the scores at each site and dividing by the number of sites evaluated. Higher scores denote higher plaque accumulation. Lower scores are more favorable.
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
units on a scale
  8wk mandibular PI score | 1.84 (0.60) | 1.77 (0.44) | 1.82 (0.46) | 1.82 (0.57)
  12wk mandibular PI score | 2.92 (0.71) | 2.93 (0.50) | 2.74 (0.52) | 2.89 (0.32)

5. Secondary Outcome: Maxillary Plaque Index (PI) Score
Description: as for outcome 4
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
units on a scale
  8wk maxillary PI score | 1.56 (0.55) | 1.71 (0.44) | 1.69 (0.49) | 1.68 (0.56)
  12 wk maxillary PI score | 2.77 (0.42) | 3 (0.32) | 2.81 (0.32) | 2.89 (0.47)

6. Secondary Outcome: Gingival Crevicular Fluid (GCF) Volume
Description: GCF will be collected by placing a filter paper strip at the opening of the gingival crevice. After carefully removing the supragingival plaque from the sampling area, a paper strip will be placed for 30s or until visibly wet. Sampling time will be recorded and GCF volume collected with each sample will be quantified using a Periotron device. GCF volume will be sampled from three mesial sites per subject: The upper left central incisor, the first upper left premolar and the first upper left molar. Should any of these teeth be missing, substitution will occur in the following order (i) the contralateral tooth, (ii) the distally adjacent tooth, or (iii) the distally adjacent tooth of the contralateral tooth. Should a sample be visibly contaminated with blood, the sample will be discarded and substitution will occur as described above.
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: ul
Arm/Group | 1-Placebo | 2-Vitamin D3, 500 IU | 3-Vitamin D3, 2500 IU | 4-Vitamin D3, 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
ul
  8wk GCF volume site 1 | 38.1 (12.5) | 49.1 (21.3) | 37.1 (10.0) | 57.6 (24.2)
  12wk GCF volume site 1 | 50.8 (13.1) | 66.5 (31.8) | 35.1 (7.8) | 55.9 (48.0)
  8wk GCF volume site 2 | 53.7 (9.8) | 53.5 (23.4) | 42.5 (27.4) | 61.0 (36.0)
  12wk GCF volume site 2 | 83.6 (24.5) | 71.9 (29.5) | 54.3 (24.6) | 72.4 (39.6)
  8wk GCF volume site 3 | 70.4 (32.9) | 92.9 (26.0) | 58.4 (19.7) | 59.9 (16.5)
  12wk GCF volume site 3 | 95.9 (27.4) | 99.1 (37.7) | 64.8 (20.0) | 92 (39.7)

7. Secondary Outcome: Gingival Crevicular Fluid (GCF) Concentrations of TNF-alpha, IL1-beta, IL-2, IL-12
Description: GCF will be collected by placing a filter paper strip at the opening of the gingival crevice. After carefully removing the supragingival plaque from the sampling area, a paper strip will be placed for 30s or until visibly wet. Sampling time will be recorded and GCF volume collected with each sample will be quantified using a Periotron device.
  GCF volume will be sampled from three mesial sites per subject: The upper left central incisor, the first upper left premolar and the first upper left molar. Should any of these teeth be missing, substitution will occur in the following order (i) the contralateral tooth, (ii) the distally adjacent tooth, or (iii) the distally adjacent tooth of the contralateral tooth. Should a sample be visibly contaminated with blood, the sample will be discarded and substitution will occur as described above. Concentrations of TNF-alpha, IL-1 beta, IL-2, and IL-12 will be measured and means and SDs will be calculated for each study arm.
Time Frame: week 8 and week 12
Measure: Mean (Standard Deviation); unit: pg/site
Arm/Group | 1-Placebo | 2-Vitamin D3, 500 IU | 3-Vitamin D3, 2500 IU | 4-Vitamin D3, 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
pg/site
  8wk TNF-alpha | 0.97 (1.14) | 1.53 (1.86) | 1.34 (1.93) | 1.87 (3.14)
  12wk TNF-alpha | 1.00 (1.04) | 1.11 (1.32) | 1.73 (3.02) | 7.94 (18.12)
  8wk IL-1 beta | 0.04 (0.00) | 0.05 (0.02) | 0.04 (0.00) | 0.04 (0.00)
  12wk IL-1 beta | 0.04 (0.00) | 0.04 (0.02) | 0.04 (0.00) | 0.04 (0.00)
  8wk IL-2 | 24.11 (34.83) | 13.44 (2.66) | 13.13 (6.52) | 13.07 (6.71)
  12wk IL-2 | 20.78 (17.31) | 12.5 (0.00) | 12.56 (0.18) | 13.36 (1.70)
  8wk IL-12 | 0.65 (1.22) | 0.11 (0.17) | 0.03 (0.04) | 0.96 (2.10)
  12wk IL-12 | 0.62 (1.10) | 0.06 (0.07) | 0.02 (0.01) | 1.08 (2.28)

8. Secondary Outcome: Serum Calcium
Description: The serum calcium blood test measures the total calcium in the participants' blood. The normal range for total serum calcium concentration in adults is 8.9-10.2 mg/dL.
Time Frame: week 7, week 12
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | 1-Placebo | 2-Vitamin D3, 500 IU | 3-Vitamin D3, 2500 IU | 4-Vitamin D3, 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
mg/dl
  7wk serum calcium | 9.6 (0.4) | 9.1 (0.3) | 9.2 (0.3) | 9.1 (0.5)
  12wk serum calcium | 9.4 (0.4) | 9.2 (0.5) | 9.2 (0.3) | 9.3 (0.2)

9. Secondary Outcome: Urinary Calcium/Creatinine Ratio
Description: Urinary calcium ratios were calculated from urine samples at week 4, 7, and 12. A normal reference interval for the urine calcium (mg/dL):urine creatinine (mg/dL) ratio is <0.14.
Time Frame: week 4, week 7, week 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 1-Placebo | 2-Vitamin D3, 500 IU | 3-Vitamin D3, 2500 IU | 4-Vitamin D3, 5000 IU
Number analyzed (Participants) | 9 | 8 | 8 | 7
ratio
  4wk calcium/creatinine ratio | 0.07 (0.1) | 0.06 (0.03) | 0.07 (0.04) | 0.09 (0.01)
  7wk calcium/creatinine ratio | 0.09 (0.1) | 0.07 (0.04) | 0.09 (0.02) | 0.13 (0.13)
  12wk calcium/creatinine ratio | 0.12 (0.1) | 0.07 (0.03) | 0.11 (0.09) | 0.11 (0.07)

ADVERSE EVENTS:
Groups:
- 2- Vitamin D3, 500 IU: vitamin D3, 500 IU capsule once per day for 12 weeks
- 3- Vitamin D3 2500 IU: vitamin D3, 2500 IU capsule once per day for 12 weeks
- 4- Vitamin D3 5000 IU: vitamin D3, 5000 IU capsule once per day for 12 weeks
Arm/Group | 1- Placebo | 2- Vitamin D3, 500 IU | 3- Vitamin D3 2500 IU | 4- Vitamin D3 5000 IU
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 1/8 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Placebo (N=9) | 2- Vitamin D3, 500 IU (N=8) | 3- Vitamin D3 2500 IU (N=8) | 4- Vitamin D3 5000 IU (N=7)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
There were recruitment delays due to the potential seasonal impact on vitamin D levels from the sun and the research center was relocated. Both resulted in lower enrollment during the funded time frame than originally projected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes